CLINICAL TRIAL: NCT00318812
Title: Heme Iron Polypeptide for the Treatment of Iron Deficiency Anemia in Pre-Dialysis Patients: A Pilot Randomized Controlled Study
Brief Title: Heme Iron Polypeptide for Iron Deficiency Anemia in Chronic Renal Failure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005840-01H
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-04

CONDITIONS: Anemia; Renal Failure
Keywords: Randomized controlled trial (RCT); Prospective Studies; ferric oxide, saccharated; Peptides; Heme; Iron; Erythropoietin,; Recombinant; Ferritin; Transferrin; Treatment Outcome
MeSH Terms: conditions — Anemia; Renal Insufficiency | interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heme Iron (Experimental): Heme Iron Polypeptide 11mg PO tid for 6 months
  Interventions: Drug: Heme Iron Polypeptide (Proferrin)
- Venofer (Active Comparator): Venofer q month IV x 6 months
  Interventions: Drug: Iron sucrose (Venofer)

INTERVENTIONS:
Drug: Heme Iron Polypeptide (Proferrin) — Heme iron polypeptide 11mg po tid for 6 months
  Other Names: Proferrin
  Arms: Heme Iron
Drug: Iron sucrose (Venofer) — Iron sucrose infusion IV q month x 6 months
  Other Names: Venofer
  Arms: Venofer

SUMMARY:
The purpose of this study is to determine if oral Heme Iron Polypeptide is as effective as intravenous (IV) iron sucrose in the treatment of iron-deficiency anemia for patients with chronic kidney disease.

DETAILED DESCRIPTION:
Iron deficiency anemia is common in patients with pre-dialysis chronic kidney disease, and is associated with significant morbidity. Conventional treatment with oral iron salts or IV iron formulations are costly and are associated with side effects. Heme iron polypeptide is a newly available formulation of oral iron which can be administered orally, is well absorbed by uremic patients, and has potentially fewer side effects.

Comparison: Iron deficient anemic patients will be randomized to either oral heme iron polypeptide or IV iron sucrose for six months.

ELIGIBILITY:
Inclusion Criteria:

* eGFR < 30 mL/min
* Hb 90-110 g/L
* Age > 18
* Not on renal replacement therapy
* Transferrin saturation < 20% OR Ferritin <100 mcg/L
* B12 & folate within reference range

Exclusion Criteria:

1. Iron overload (Tsat > 50% or ferritin > 800 μg/L);
2. malignancy; recurrent gastro-intestinal bleeding, major surgery or infection within the last 3 months;
3. parenteral iron therapy, blood transfusion within the last 3 months;
4. pregnancy;
5. contraindication to any study medication and;
6. inability or refusal to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Zimmerman, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Nagaraju SP, Cohn A, Akbari A, Davis JL, Zimmerman DL. Heme iron polypeptide for the treatment of iron deficiency anemia in non-dialysis chronic kidney disease patients: a randomized controlled trial. BMC Nephrol. 2013 Mar 20;14:64. doi: 10.1186/1471-2369-14-64. PMID 23514036

RESULTS

PARTICIPANT FLOW:
Recruitment Details: May 2007 - February 2011, 55 Chronic Kidney Disease patients >18years,with an estimated Glomerular Filtration Rate (eGFR) <30mls/minute and Hemoglobin (Hgb) of 90-110 were recruited. Recruitment was expanded to eGFR ≤60 and Hgb of 90-120g/L (females)and 90-135 g/L (males) with serum ferritin < 100 mcg /L or Transferrin Saturation (TSAT) < 20%)
Pre-assignment Details: 15 of the 55 patients were screen failures due to; Hgb too high/low, ferritin level too high, Vitamin B level too low,one had bypass surgery
Groups:
- Iron Sucrose: Iron Sucrose q month IV x 6 months
Period: Overall Study
Arm/Group | Heme Iron | Iron Sucrose
Started | 18 | 22
Completed | 18 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Heme Iron | Iron Sucrose | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 76 [66 to 83] | 66 [58 to 76] | 68 [63 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 13 | 12 | 25
Region of Enrollment [Number; unit: participants]
  Canada | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin Concentration at 6 Months
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | Heme Iron | Iron Sucrose
Number analyzed (Participants) | 18 | 22
g/L | 117 [110 to 129] | 113 [108 to 120]

2. Secondary Outcome: Ferritin
Description: Comparison of Ferritin at 6 months between the 2 Groups
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: ug/L
Arm/Group | Heme Iron | Iron Sucrose
Number analyzed (Participants) | 18 | 22
ug/L | 85.5 [44 to 104] | 244 [72 to 298]

3. Secondary Outcome: Transferrin Saturation
Description: Comparison of Transferrin Saturation between the Groups
Time Frame: 6 Months
Measure: Median (Inter-Quartile Range); unit: percentage of bound iron sites
Arm/Group | Heme Iron | Iron Sucrose
Number analyzed (Participants) | 18 | 22
percentage of bound iron sites | 21.5 [17 to 29] | 21.5 [17 to 27]

ADVERSE EVENTS:
Arm/Group | Heme Iron | Iron Sucrose
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 5/18 | 4/22
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heme Iron (N=18) | Iron Sucrose (N=22)
constipation (Gastrointestinal disorders) | 5 (5) | 4 (4) — Gastrointestinal complaints were the most common adverse effects in both groups with constipation and abdominal cramps being the most common in HIP group and constipation in IV sucrose group
abdominal cramps (Gastrointestinal disorders) | 5 (5) | 3 (3)
Symptomatic Hypotension (Cardiac disorders) | 0 (0) | 3 (3) — symptomatic hypotesnion was seen in 3 patients in the IV sucrose arm and 0 patients in the HIP arm
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)

LIMITATIONS AND CAVEATS:
Recruitment for the trial was a challenge; over 1100 patients screened - 55 consented - 40 randomized

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No